CLINICAL TRIAL: NCT01788878
Title: Cancer of the Upper Aero-digestive Tract and Socio-professional Future
Acronym: CARDEL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Oscar Lambret (Other)
Collaborators: University Lille 3 (Unknown); Région Nord-Pas de Calais, France (Other); University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CARDEL-1211
Record Dates: First submitted 2013-01-31; First posted 2013-02-11 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Upper Aerodigestive Tract Neoplasms
Keywords: socio-professional future
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Questionnaires (Experimental): completion of questionnaires
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Questionnaires — A first series of questionnaires will be given by the investigator at patients before treatment (inclusion visit) and then the questionnaires will be given at the follow-up visits planned at 6 months, 12 months and 18 months.
  Medical data will be collected via the CRF.

SUMMARY:
The aim of this study is to explore the main factors associated with the return to work of patients presenting an upper aero-digestive tract cancer.

DETAILED DESCRIPTION:
Socio-professional, medical, psychological, demographic, economic, and educational data collection in patients within the care pathway of upper aero-digestive tract cancer.

A series of questionnaires will be presented at the initial consultation and then at 6 months, at 12 months and at 18 months during follow-up visits. Medical data will be collected via the CRF.

ELIGIBILITY:
Inclusion Criteria:

* Age at diagnosis ≥ 18 to ≤ 55 years
* Employed at the entry into the care pathway
* Presenting an upper aero-digestive tract cancer (excluding nasal cavities), stage I, II and III, under a first anti-tumor treatment (surgery, radiotherapy, or chemotherapy)
* Patient mastering the French language
* Affiliated to the social security system
* Consent signed by the patient before the implementation of any specific study procedure

Exclusion Criteria:

* Having been treated for another cancer before (except skin cancer and / or prostate)
* Metastatic disease from the outset
* Patient unable to submit to a regular follow-up
* Presenting psychiatric disorders

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2014-02; Primary Completion 2016-08 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Main psycho-medical and socio-professional determinants associated with return to work at 18 months after diagnosis | At month 18

SECONDARY OUTCOMES:
Period until return to work (also part-time work) | At month 6, month 12, month 18
Modalities, period and stability of this return to work | At month 6, month 12, month 18
Alternatives to return to work (retirement, disability, etc ...) | At month 6, month 12, month 18
Psychological factors that might interfere with the behaviors to return to work | At baseline, Month 6, Month 12, Month 18
Information collected in the perceived support part of the questionnaire | At baseline, Month 6, Month 12, Month 18

CONTACTS AND LOCATIONS:
Overall Officials: Sophie FANTONI, Pr, Study Director — CHRU de Lille; Jean-Louis LEFEBVRE, Pr, Study Director — Centre Oscar Lambret
Locations (8):
- France (8):
  - CHU de Caen, Caen
  - Centre François Baclesse, Caen
  - Hôpital privé de l'Estuaire, Le Havre
  - Centre Oscar Lambret, Lille
  - CHRU de Lille, Lille
  - Hôpital de la Timone, Marseille
  - Centre Antoine Lacassagne, Nice
  - CHU de Rouen, Rouen

IPD SHARING:
Plan to Share IPD: No